CLINICAL TRIAL: NCT06322290
Title: Epidemiological Study on Invasive Bacterial Diseases (IBD)
Brief Title: Epidemiological Study on Invasive Bacterial Diseases
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Chiara Azzari, Full professor, Meyer Children's Hospital IRCCS
Other Study IDs: SEMBAI
Record Dates: First submitted 2024-02-28; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Invasive Bacterial Diseases (IBD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for bacterial identification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pneumococcal, meningococcal, and hemophilus Invasive Bacterial Diseases: Pediatric and adult patients diagnosed with pneumococcal, meningococcal, and hemophilus Invasive Bacterial Diseases, as defined in the Italian Superior Institute of Health (ISS) protocol.
  Interventions: Diagnostic Test: assessment of pathogens in blood specimens

INTERVENTIONS:
Diagnostic Test: assessment of pathogens in blood specimens — Molecular diagnosis of Invasive bacterial diseases due to Streptococcus pneumoniae, Neisseria meningitidis and Haemophilus influenzae

SUMMARY:
Streptococcus pneumoniae (pneumococcus), Neisseria meningitidis (meningococcus), and Haemophilus influenzae (hemophilus) are among the main bacteria responsible for invasive bacterial diseases (MBIs) that result in severe clinical pictures also characterized by a high frequency of serious complications. Surveillance of infections caused by these pathogens and their distribution by serotypes/serogroups is essential to guide public health interventions, assess epidemiologic trends, monitor any secondary cases, estimate the proportion of preventable cases, identify any vaccine failures, and evaluate the impact of vaccine strategies.The present study aims to study the epidemiology of invasive bacterial diseases, characterize the circulating strains also in order to plan treatment and prevention strategies.

DETAILED DESCRIPTION:
Pathogen identification by culture methods has been shown to be unsatisfactory, as antibiotic therapy carried out in patients before hospitalization prevents bacterial culture development and subsequent typing in many cases. In addition, technical problems due to sample collection, storage and transport reduce germ viability leading to false negatives in pathogen identification by culture methods. In contrast, molecular diagnosis allows germ identification on biological samples even in the absence of germ viability, thus enabling more accurate diagnosis.

Surveillance of infections caused by these pathogens and their distribution by serotypes/serogroups is essential to guide public health interventions, assess epidemiological trends, monitor any secondary cases, estimate the proportion of preventable cases, identify any vaccine failures, and evaluate the impact of vaccine strategies.In 2006, the AOU Meyer Immunology Laboratory received a grant from the National Center for Disease Prevention and Control (NCDC) to develop a molecular diagnostic method for surveillance of invasive infections with Neisseria meningitidis (meningococcal,) Streptococcus pneumoniae (pneumococcus) and Haemophilus influenzae (hemophilus) that would allow identification of the germ on biological samples even in the absence of germ viability, with a view to improving surveillance, prevention and treatment strategies. The project involved performing molecular diagnostic tests on samples from patients referred to hospitals in the Tuscany Region and outside the region. The present study aims to study the epidemiology of invasive bacterial diseases, characterize the circulating strains also in order to plan treatment and prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adult patients diagnosed with pneumococcal, meningococcal, and hemophilus MBI

Exclusion Criteria:

* Other type of bacterial infections.

Ages: 1 Day to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients diagnosed with pneumococcal, meningococcal, and hemophilus Infective bacterial disease in Italy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2031-12-30 (Estimated); Study Completion 2032-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Infective Bacterial Diseases from Streptococcus pneumoniae (pneumococcus) during the study period in pediatric age. | Through study completion, an average of 1 year
  Monitor the trend of Infective Bacterial Diseases cases Streptococcus pneumoniae (pneumococcus) in Italy, during pediatric age.
Incidence rate of of Infective Bacterial Diseases cases from Neisseria meningitidis during the study period in pediatric age. | Through study completion, an average of 1 year
  Frequencies of Infective Bacterial Diseases cases from Neisseria meningitidis in Italy (meningococcus)
Incidence rate of Infective Bacterial Diseases cases from Haemophilus influenzae during the study period in pediatric age. | Through study completion, an average of 1 year
  Frequencies of Infective Bacterial Diseases cases from Haemophilus influenzae (hemophilus) in Italy

SECONDARY OUTCOMES:
Frequency of circulating serogroups/serotypes in Italy for S.pneumoniae, N.meningitidis, H.influenzae. | Through study completion, an average of 1 year
  Describe the distribution of circulating serogroups/serotypes
Proportion of these invasive infections (S.pneumoniae, N.meningitidis, H.influenzae) that are preventable by vaccine in Italy | Through study completion, an average of 1 yeary
  Estimate the proportion of these invasive infections that are preventable by vaccine
Vaccine failure rate for S.pneumoniae, N.meningitidis, and H.influenzae. | Through study completion, an average of 1 year
  Assessing rate cases of vaccine failure

CONTACTS AND LOCATIONS:
Locations (38):
- Italy (38):
  - Ospedale di Adria, Adria
  - Ospedali riuniti di Ancona, Ancona
  - Ospedale di Andria, Andria
  - Ospedale Giovanni XXIII, Bari
  - Policlinico S.Orsola-Malpighi IRCCS, Bologna
  - Fondazione poliambulanza Brescia, Brescia
  - Ospedale Giovanni XXIII, Brescia
  - Ospedale di Campobasso, Campobasso
  - Ospedale Camposampiero, Camposampiero
  - Ospedale di Esine asst Valcamonica, Esine
  - Ospedale di Feltre (AULSS 1 Dolomiti), Feltre
  - Immunology Laboratory Meyer Children's Hospital IRCCS, Florence
  - Ospedale Morgagni, Forlì
  - AO Salvini di Garbagnate, Garbagnate
  - Azienda sanitaria universitaria Giuliano Isontina (ASU GI), Gorizia
  - Ospedale di Macerata, Macerata
  - Ospedale di Magenta, Magenta
  - Azienda Ospedaliera Policlinico Universitario "G. Martino", Messina
  - IRCCS San Raffaele, Milan
  - AORN Santobono, Napoli
  - AOU Federico II di Napoli, Napoli
  - Ospedale di Novara, Novara
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Ospedale spirito santo di Pescara, Pescara
  - Azienda sanitaria Friuli occidentale, Pordenone
  - Ospedale degli infermi, Rimini
  - Ospedale Pediatrico Bambin Gesù IRCCS, Roma
  - Ospedale Sandro Pertini, Roma
  - Ospedale San Leonardo di Salerno, Salerno
  - Ospedale di Saronno, Saronno
  - AOU Sassari, Sassari
  - Ospedale di Scorrano, Scorrano
  - ASP Trapani, Trapani
  - IRCCS Materno Infantile Burlo Garofolo, Trieste
  - Azienda sanitaria universitaria Friuli Centrale (ASU FC), Udine
  - Azienda ospedaliera universitaria integrata Verona, Verona
  - Ospedale civile di Vibo Valentia, Vibo Valentia
  - Ospedale Maggiore Carlo Alberto Pizzardi, Bologna, Ì

IPD SHARING:
Plan to Share IPD: No